CLINICAL TRIAL: NCT04085848
Title: A Controlled, Randomized Study Evaluating the Effecacy of Receptive Music Therapy on Psychological Pain in Suicidal Patients
Brief Title: Music Against Psychological Pain in Suicide
Acronym: MAPPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017/CHU/19
Record Dates: First submitted 2019-09-03; First posted 2019-09-11 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Suicide, Attempted; Suicidal Ideation
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Groupe intervention (Experimental): Usual care and music therapy
  Interventions: Other: music therapy
- Groupe contrôle (No Intervention): Usual care

INTERVENTIONS:
Other: music therapy — 4 music therapy sessions during a period of time of 48 hours. Each session lasts 30 minutes.
  Arms: Groupe intervention

SUMMARY:
This study compares the efficacy of music therapy associated with standard care versus the standard care alone on the psychological pain in suicidal patients.

DETAILED DESCRIPTION:
Music therapy consists of using the Music Care tool. Each patient randomized in the music therapy arm should perform 4 music therapy sessions of 30 minutes on 48h.

Before and after each music therapy sessions, the psychological pain will be measured by the analogical visual scale.

Standard care consists of a medical and paramedical interview lasting 20-30 minutes. At the end of the interview, a drug treatment (BZD anxiolytic and/or hypnotic) is prescribed and the patient is hospitalized. During hospitalization, patient is regularly interviewed in order to evaluate his psychological status.

ELIGIBILITY:
Inclusion Criteria:

* Patient with suicidal ideas, thoughts or surviving suicide attempt
* Patient whose emergency somatic management lasted less than 48h
* Patient who, according to the physician, is still in suicidal mood
* Patient admitted in the psychiatric hospitalization unit of the Public Mental Health Establishment
* Patient with voluntary admission and agrees to stay in hospital from 48h to 60h
* Patient able to write and read in french
* Patient affiliated to a social security scheme
* Patient who gives his Informed consent before any procedure related to the study

Exclusion Criteria:

* Patient with attempt suicide requiring a somatic care (intensive, surgery, gastric lavage...)
* Patient with medical history of audiogenic and/or musicogenic epilepsy
* Patient with major impairment of hearing function
* Patient unable to support the headhset earphone
* Patient with contra indication to BZD, hypnotics (Zopiclone) or requiring more sedative and/or psychotic drugs
* Patient under guardianship or under judicial protection
* Patient hospitalized at the request of a third party or ex officio

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from inclusion psychological pain at 48 hours after inclusion | 48 hours after inclusion
  Pain analogical visual scale (scale ranges : from 0 to 10) min = 0 = no psychological pain and max = 10 = maximum psychological pain

CONTACTS AND LOCATIONS:
Overall Officials: Erick GOKALSING, Principal Investigator — EPSMR
Locations (1):
- Etablissement Public de Santé Mentale de La Réunion, Saint-Paul, Reunion

IPD SHARING:
Plan to Share IPD: No